CLINICAL TRIAL: NCT06817226
Title: Cultural and Linguistic Adaptation of a Breast Reconstruction Decision Tool - AIM2
Brief Title: BREAST Choice Decision Tool R21 - AIM2
Acronym: BREASTChoice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-1340 - AIM2; R21CA287321 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Surgery; Breast reconstruction; mastectomy; Spanish-speaking; Latina; The BREASTChoice
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer survivors (Other): Latina breast cancer survivors.
  Interventions: Behavioral: Pre-survey; Behavioral: BREASTChoice tool.; Behavioral: Post-survey

INTERVENTIONS:
Behavioral: Pre-survey — Participants will take a pre-survey to measure demographics, health literacy, numeracy and breast reconstruction decision quality.
Behavioral: BREASTChoice tool. — Participants will then engage in a self-guided review of the adapted BREASTChoice tool.
Behavioral: Post-survey — Participants will take the post-survey to assess breast reconstruction decision quality.

SUMMARY:
Breast reconstruction is a critical component of breast cancer treatment because it restores quality of life and body image after mastectomy. However, Spanish-speaking Latina women are significantly less likely to undergo reconstruction (13.5% vs. 41% for non-Latina White or highly acculturated Latina), meet with a reconstructive surgeon (18.1% vs. 72.6% for non-Latina White), or receive adequate information. Spanish-speaking Latina breast cancer survivors who do not have reconstruction experience the highest rates of decisional dissatisfaction and regret, compared to any other group of breast cancer survivors.

Persons diagnosed with cancer who primarily speak Spanish and identify as Latin American (hereafter we use the term "Spanish-speaking Latinx/a cancer survivor") are less likely to receive guideline-concordant treatment and more likely to have poor cancer outcomes. One way to improve guideline-concordant treatment is through shared decision-making and decision support. When a decision is preference-sensitive (the right choice depends on the person's preferences), such as decisions about breast reconstruction after mastectomy, decision aids are effective. Unfortunately, most decision aids in the United States are written in English and developed or tested with few Latinx people.

The BREASTChoice decision aid, proven effective in two randomized controlled trials, addresses knowledge gaps in breast cancer survivors. This study focuses on developing a Spanish-language version of BREASTChoice, which was previously unavailable. For that reason, the Cultural and Linguistic Adaptation Framework (CLAF) incorporates qualitative and experiential data to adapt BREASTChoice. The adaptation process takes place in five steps: appraise, review, assess, solicit, and integrate.

ELIGIBILITY:
Inclusion Criteria for Survivors: (must meet all criteria)

* Female sex
* Adult at least 18 years of age
* Latina, Latino, or Latinx ethnicity - defined as born in or descending from South America, Mexico, Central America, other Spanish-speaking Caribbean islands
* Prefer to receive health information in Spanish
* Have a history of breast malignancy (e.g., ductal carcinoma, DCIS) or high risk for breast cancer (e.g., BRCA mutation)
* Had breast surgery (Mastectomy/Lumpectomy/Mastectomy but no reconstruction) within the last 8 years
* Able to understand an IRB-Approved consent information sheet

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Change in breast reconstruction knowledge | Up to 2 months
  Knowledge will be calculated before and after the intervention. The number of correct answers divided by the total number of knowledge items. Missing items will be counted as incorrect. A knowledge score will be calculated only if at least 50% of the items are answered. Descriptive statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Lee, MPP, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- The University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials